CLINICAL TRIAL: NCT06430515
Title: The Clinical Efficacy and Safety of Intratumoral Injection of Chemotherapy for Advanced Solid Tumors Through Fine Needle Puncture
Brief Title: The Clinical Efficacy and Safety of Intratumoral Injection of Chemotherapy for Advanced Solid Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY23197
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Intratumoral Injection; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intratumoral Injection of Chemotherapy (Experimental): Fine-needle puncture guided by CT or ultrasound and infusion of chemotherapeutic agents (e.g. cisplatin, oxaliplatin, etc.) via the tumour increases the local drug concentration in the tumour, improves therapeutic efficacy and reduces drug resistance and systemic adverse effects.
  Interventions: Procedure: Intratumoral Injection of Chemotherapy

INTERVENTIONS:
Procedure: Intratumoral Injection of Chemotherapy — This project intends to investigate the clinical efficacy of intra-tumoural injection of chemotherapeutic agents (e.g. cisplatin, oxaliplatin, etc.)via fine needle aspiration guided by CT or ultrasound in patients with advanced solid cancers to validate the safety and efficacy.

SUMMARY:
This project intends to investigate the clinical efficacy of intra-tumoural injection of chemotherapeutic agents (e.g. cisplatin, oxaliplatin, etc.)via fine needle aspiration guided by CT or ultrasound in patients with advanced solid cancers to validate the safety and efficacy.

DETAILED DESCRIPTION:
Malignant solid tumours including lung and liver cancers are the most common malignant tumours worldwide and have a very high mortality rate. Currently,the clinical practice mainly relies on systemic administration of chemotherapeutic agents usually by intravenous infusion for patients with solid cancer with multiple metastases,but the overall efficiency is not high.Single or multiple chemotherapeutic agents are infused intratumourally to increase the local drug concentration in the tumour, improve efficacy and reduce drug resistance and systemic adverse effects. This project intends to investigate the clinical efficacy of intra-tumoural injection of chemotherapeutic agents (e.g. cisplatin, oxaliplatin, etc.)via fine needle aspiration guided by CT or ultrasound in patients with advanced solid cancers to validate the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18-75 years;
2. Subjects must have histologically- or cytologically-confirmed diagnosis of advanced solid tumor(s) and have progressed on or is not eligible for available standard therapy;
3. Subjects have at least one measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (non-nodal lesions with longest diameter ≥ 10 mm, or nodal lesions with short diameter ≥ 15 mm);
4. ECOG score of 0-2, lifespan > 12 weeks;
5. Women of childbearing age who have a negative pregnancy test within 7 days before treatment. Female patients of childbearing age, and male patients with partners of childbearing age must agree to use at least one medically recognized contraceptive method during study treatment and within at least 6 months after the last dose of investigational drug;
6. Voluntarily participated in this study, signed the informed consent form, had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. The patient is diagnosed with central nervous system leukemia(symptoms, signs, imaging, cerebrospinal fluid);
2. White blood cell count ≥ 50×10^9/ L or patients with rapid disease progression can't be guaranteed to complete a full treatment cycle;
3. Patients with fungal, bacterial, viral or other uncontrollable infections or requiring four-level isolation treatment.
4. HIV, HBV and HCV positive;
5. Patients with diseases of the central nervous system or autoimmune central nervous system lesions, Including stroke, epilepsy, dementia;
6. Patients have myocardial infection, cardiac angiography or stents, active angina or other obvious clinical symptoms, or have cardiopathic asthma or cardiovascular lymphocytic infiltrates，within 12 months;
7. Patients are on anticoagulation or have severe coagulopathy (APTT>70);
8. Patients in any condition requiring systemic treatment with corticosteroids or other immunosuppressive agents within 2weeks prior to investigational drug administration;
9. Subjects having any serious uncontrolled disease or in other conditions that would preclude them from receiving study treatment and are considered unsuitable for this study in the opinion of the investigator;
10. Subjects in other conditions that are considered unsuitable for this study by the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Relief degree of tumors | through study completion, an average of 5 year
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST1.1）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 3 years, year 3
  The duration from the beginning of treatment to cancer recurrence or progression
Overall survival（OS） | 5 years, year 5
  The duration from the beginning of treatment to patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China